CLINICAL TRIAL: NCT02595502
Title: Clinical Evaluation of Two Silicone Hydrogel Daily Disposable Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CR-5743
Record Dates: First submitted 2015-11-02; First posted 2015-11-03 (Estimated); Results first posted 2016-07-20 (Estimated); Last update posted 2017-07-05 (Actual); Status verified 2017-06

CONDITIONS: Vision Disorders
MeSH Terms: conditions — Vision Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sequence 1: Test Control Test (Active Comparator): Test/control/test using the Johnson & Johnson Vision Care (JJVC) Marketed contact lens (test) and the Competitor Marketed contact lens (control). Lenses will be worn as daily wear, daily disposable on both eyes for approximately one week each in between lenses for total study duration of approximately three weeks per subject. Subjects are required to wear the lenses at least five days for at least eight hours per day worn.
  Interventions: Device: JJVC Marketed Contact Lens (Test); Device: Competitor Marketed Contact Lens (Control)
- Sequence 2: Control Test Control (Active Comparator): Control/test/control using the JJVC Marketed contact lens (test) and the Competitor Marketed contact lens (control). Lenses will be worn as daily wear, daily disposable on both eyes for approximately one week each for total study duration of approximately three weeks per subject. Subjects are required to wear the lenses at least five days for at least eight hours per day worn.
  Interventions: Device: JJVC Marketed Contact Lens (Test); Device: Competitor Marketed Contact Lens (Control)

INTERVENTIONS:
Device: JJVC Marketed Contact Lens (Test)
  Other Names: senofilcon A
Device: Competitor Marketed Contact Lens (Control)
  Other Names: delefilcon A

SUMMARY:
The purpose of this investigation is to evaluate the short-term, clinical performance of two silicone hydrogel daily disposable contact lenses.

ELIGIBILITY:
Inclusion Criteria:

* The subject must read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
* The subject must appear able and willing to adhere to the instructions set forth in this clinical protocol.
* The subject must be between (and including) 18 and 39 years of age.
* The subject must be an adapted wearer of spherical soft contact lenses in both eyes. That is, the subject must wear their habitual lenses at least five (5) days per week and eight (8) hours per day worn for at least 30 days immediately preceding the study.
* The subject must have vertex-corrected distance refraction that allows a plano over-refraction with the available contact lens powers of -0.50 to -6.00 Diopters (D) in each eye.
* The subject must have refractive astigmatism, if present, of less than or equal to 1.00 D in each eye.
* The subject must have best corrected visual acuity of 20/25 or better in each eye.

Exclusion Criteria:

* Currently pregnant or breastfeeding (subjects who become pregnant during the study will be discontinued).
* Any ocular or systemic allergies or diseases that may interfere with contact lens wear.
* Any autoimmune disease or use of medication, which may interfere with contact lens wear.
* Entropion, ectropion, extrusions, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, or aphakia.
* Any previous, or planned, ocular or interocular surgery (e.g., radial keratotomy, photorefractive keratectomy (PRK), laser-assisted in situ keratomileusis (LASIK), etc.).
* Any grade 3 or greater slit lamp findings (e.g., edema, corneal neovascularization, corneal staining, tarsal abnormalities, conjunctival injection) on the FDA classification scale, any previous history or signs of a contact lens-related corneal inflammatory event (e.g., past peripheral ulcer or round peripheral scar), or any other ocular abnormality that may contraindicate contact lens wear.
* Any ocular infection.
* Any corneal distortion resulting from previous hard or rigid gas permeable contact lens wear.
* Monovision, multi-focal, toric, or extended wear contact lens correction.
* Participation in any contact lens or lens care product clinical trial within 14 days prior to study enrollment.
* History of binocular vision abnormality or strabismus that is likely to affect successful contact lens wear.
* Any infectious disease (e.g., hepatitis, tuberculosis) or contagious immunosuppressive diseases (e.g., HIV) by self-report.

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 286 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2015-11-01 (Actual); Study Completion 2015-11-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - Becky Bizzle, OD, Montgomery, Alabama
  - Complete Family Eye Care of Fruit Cove, Fruit Cove, Florida
  - Golden Family Eyecare, Sarasota, Florida
  - St. Lucy's Vision Center, Tampa, Florida
  - Eye Associates of Winter Park, Winter Park, Florida
  - VisualEyes, Inc., Roswell, Georgia
  - Advantage Eyecare Associates, LLC, Neodesha, Kansas
  - Sacco Eye Group, Vestal, New York
  - Advanced Family Eye Care, Denver, North Carolina
  - total Eye Care PA, Memphis, Tennessee
  - Brian Frazier, OD, Jacksonville, Texas
  - Timothy R. Poling, OD, Roanoke, Virginia
  - Ziegler Leffingwell Eyecare, West Allis, Wisconsin

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 286 subjects were enrolled in this study. Of the enrolled subjects 1 subject did meet the eligibility criteria and 285 subjects were randomized. Of the randomized subjects 9 were discontinued and 276 completed the study.
Groups:
- Delefilcon A /Senofilcon A/Delefilcon A: Subjects that wore the delefilcon A lens first, the senofilcon A lens second and then wore the delefilcon A lens again, third.
- Senofilcon A/Delefilcon A/Senofilcon A: Subjects that wore the senofilcon A lens first, the delefilcon A lens second and then wore the senofilcon A lens again, third.
Period: Period 1
Arm/Group | Delefilcon A /Senofilcon A/Delefilcon A | Senofilcon A/Delefilcon A/Senofilcon A
Started | 143 | 142
Completed | 142 | 140
Not Completed | 1 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 0 | 1
Period: Period 2
Arm/Group | Delefilcon A /Senofilcon A/Delefilcon A | Senofilcon A/Delefilcon A/Senofilcon A
Started | 142 | 140
Completed | 141 | 138
Not Completed | 1 | 2
Not completed — Adverse Event | 1 | 1
Not completed — Received incorrect lens at Period 1 | 0 | 1
Period: Period 3
Arm/Group | Delefilcon A /Senofilcon A/Delefilcon A | Senofilcon A/Delefilcon A/Senofilcon A
Started | 141 | 138
Completed | 140 | 136
Not Completed | 1 | 2
Not completed — Protocol Violation | 0 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Received Incorrect Treatment at period 3 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All subjects that were dispensed at least one study lens.
Groups:
- Dispensed Subjects: All subjects that were dispensed at least one study lens throughout the duration of the study.
Arm/Group | Dispensed Subjects
Number analyzed (Participants) | 285
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.1 (6.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 198
  Male | 87
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 3
  Asian | 6
  Black or African American | 36
  White | 238
  Other | 2
Region of Enrollment [Number; unit: participants]
  United States | 285

OUTCOME MEASURES:

1. Primary Outcome: Overall Comfort
Description: Overall comfort was assessed using the Contact Lens User Experience™ (CLUE) questionnaire. CLUE is a validated patient-reported outcomes (PRO) questionnaire to assess patient-experience attributes of soft contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Derived CLUE scores using Item Response Theory (IRT) follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response with a range of 0-120. Please note this was a 2 treatment by 3 period study design. Therefore, some subjects were randomized to receive one of the study lenses twice, hence the number of observations were summarized per lens type. For the senofilcon A lens 134+138+134=406 (Observations- 1 per subject per period, however 1 observation was not recorded) from period 1, 2 and 3 respectively. For the delefilcon A lens 138+134+138=410 from period 1, 2 and 3 respectively.
Time Frame: 1 Week
Population: The analysis population consists of subjects that completed the study without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Number of Observations
Groups:
- Delefilcon A: Subjects that wore the delefilcon A lens in any of the 3 periods during the course of this study.
- Senofilcon A: Subjects that wore the senofilcon A lens in any of the 3 periods during the course of this study.
Arm/Group | Delefilcon A | Senofilcon A
Number analyzed (Participants) | 272 | 272
Number analyzed (Number of Observations) | 410 | 405
units on a scale | 63.07 (27.752) | 71.87 (26.494)

ADVERSE EVENTS:
Time Frame: Throughout the duration of the study. Approximately 3 months.
Arm/Group | Delefilcon A | Senofilcon A
Serious Adverse Events (participants affected / at risk) | 0/285 | 0/285
Other Adverse Events (participants affected / at risk) | 0/285 | 0/285

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days